CLINICAL TRIAL: NCT04609826
Title: A Phase 1, FIH, Dose Escalation Study of JNJ-74856665 (Dihydroorotate Dehydrogenase [DHODH] Inhibitor) Alone or in Combination in Participants With AML or MDS
Brief Title: A Study of JNJ-74856665 in Participants With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Acronym: DHODH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108874; 74856665AML1001 (Other: Janssen Research & Development, LLC); 2020-002375-35 (EudraCT Number); 2024-513918-35-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: JNJ-74856665 (Experimental): Participants will receive JNJ-74856665 orally in a 21-day cycle. The dose levels will be escalated based on the decisions of the Study Evaluation Team (SET) until a recommended Phase 2 dose (RP2D) has been identified.
  Interventions: Drug: JNJ-74856665
- Arm B: JNJ-74856665 + Azacitidine (AZA) (Experimental): Participants will receive JNJ-74856665 orally in combination with AZA administered intravenously (IV) or subcutaneously (SC) in a 28-day cycle.
  Interventions: Drug: JNJ-74856665; Drug: AZA
- Arm C: JNJ-74856665 + Venetoclax (VEN) (Experimental): Participants will receive JNJ-74856665 orally in combination with VEN in a 28-day cycle.
  Interventions: Drug: JNJ-74856665; Drug: VEN
- Arm D: JNJ-74856665 (Experimental): Participants will receive JNJ-74856665 orally in a 21-day cycle. Participants with transfusion dependent relapsed/refractory Myelodysplastic Syndrome (MDS) will be included.
  Interventions: Drug: JNJ-74856665

INTERVENTIONS:
Drug: JNJ-74856665 — JNJ-74856665 will be administered orally.
Drug: AZA — AZA will be administered IV infusion or SC injection.
  Arms: Arm B: JNJ-74856665 + Azacitidine (AZA)
Drug: VEN — VEN tablet will be administered orally.
  Arms: Arm C: JNJ-74856665 + Venetoclax (VEN)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, maximum tolerated doses (MTDs) and recommended Phase 2 doses (RP2Ds) of JNJ-74856665 as monotherapy and/or in combinations.

DETAILED DESCRIPTION:
This is first-in-human (FIH) Phase 1, dose escalation study of JNJ-74856665 alone or in combination with Azacitidine or Venetoclax in participants with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS). Participants with Chronic Myelomonocytic Leukemia (CMML) are also eligible and will either receive JNJ-74856665 as monotherapy or in combination with Azacitidine. AML is a heterogeneous disease characterized by uncontrolled clonal expansion of hematopoietic progenitor cells (myeloid blasts) in the peripheral blood, bone marrow, and other tissues and is the second most common form of leukemia. MDS are a heterogeneous group of malignant hematopoietic stem cell disorders that are characterized by cytopenias, myeloid dysplasia, and a risk of transformation to AML. JNJ-74856665 is an orally bioavailable, potent, and selective dihydroorotate dehydrogenase (DHODH) inhibitor that binds to the enzyme's ubiquinone binding site promoting AML/MDS differentiation as well as cell cycle arrest and apoptosis. Azacitidine (5-azacytidine) is a nucleoside metabolic inhibitor that has been US Food and Drug Administration-approved for several MDS subtypes. Venetoclax (VEN) is a BCL-2 inhibitor that can restore activation of apoptosis in malignant cells, the survival of which often depends on dysregulation of this pathway. The study is divided into 3 periods: a Screening Phase (within 28 days before the first dose of study drug), a Treatment Phase (first dose of study drug until the completion of the end-of-treatment visit) and a Post-treatment Follow-up Phase (up to the end of study participation or end of study). The end of study is defined as the last study assessment for the last participant in the study. Total duration of study is up to 2 years and 10 months. Efficacy, safety, pharmacokinetics (PK), and biomarkers will be assessed at specified time points during this study. Participants safety and study conduct will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of: Arms A and C: Acute Myeloid Leukemia (AML) according to the World Health Organization (WHO) 2016 criteria with relapsed or refractory disease and have exhausted or are ineligible for standard therapeutic options; or newly transformed secondary AML according to the WHO 2016 criteria and have exhausted standard therapeutic options for AML during their treatment prior to transformation; or high-risk or very high-risk Myelodysplastic Syndrome (MDS) according to the WHO 2016 criteria and the revised International Prognostic Scoring System (IPSS-R) with relapsed or refractory disease and have exhausted or are ineligible for standard therapeutic options; or Arm A only: chronic myelomonocytic leukemia-2 (CMML-2) according to the WHO 2016 criteria with relapsed or refractory disease and have exhausted or are ineligible for standard therapeutic options; Arm B: Eligible participants must be considered unsuitable for intensive treatment with a curative intent (including stem cell transplantation), but eligible to receive Azacitidine (AZA) treatment with the following underlying diseases: AML (newly diagnosed or relapsed/refractory) according to the 2016 WHO classification only if Venetoclax (VEN) + hypomethylating agent (HMA) (or low-dose cytarabine) is not indicated or available; or high-risk or very high-risk MDS according to the 2016 WHO classification and IPSS-R; or CMML-2 according to the WHO 2016 criteria; Arm D: Very low, low, or intermediate-risk MDS according to the 2016 WHO classification and IPSS-R and the following: Transfusion dependence defined as requiring at least 3 red blood cell (RBC) units transfused within 16 weeks prior to C1D1; pre-transfusion hemoglobin (Hb) should be less than (<) 9.0 grams per decilitre (g/dL) to count towards the 3 units total, Relapsed/refractory to erythropoiesis-stimulating agent (ESA) treatment or endogenous serum erythropoietin (EPO) level greater than (>) 500 milliunits per milliliter (mU/mL). Exception: Del(5q) karyotype is allowed, provided prior treatment with lenalidomide has failed or participant was ineligible to receive lenalidomide
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Women of childbearing potential (WOCBP) must have a negative highly sensitive serum (beta-human chorionic gonadotropin) at screening and again within 48 hours prior to the first dose of study treatment. A urine or serum test is acceptable at subsequent time points
* A WOCBP must agree to all the following during the study and for 6 months after the last dose of study treatment: a) use a barrier method of contraception; b) use a highly effective preferably user-independent method of contraception; c) not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction; d) not plan to become pregnant; e) not breast-feeding
* A male must agree to all the following during the study and for 90 days after the last dose of study treatment: a) wear a condom when engaging in any activity that allows for passage of ejaculate to another person; b) not to donate sperm or freeze for future use for the purpose of reproduction; c) not plan to father a child. In addition, the participant should be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak

Exclusion Criteria:

* Acute promyelocytic leukemia according to World Health Organization 2016 criteria
* Known central nervous system involvement
* Prior treatment with a dihydroorotate dehydrogenase (DHODH) inhibitor for an oncology indication or intolerance to a DHODH inhibitor given for non-oncology indication
* Toxicities (except for alopecia, peripheral neuropathy, thrombocytopenia, neutropenia, anemia) from previous anticancer therapies that have not resolved to baseline or to Grade 1 or less
* Known allergies, hypersensitivity, or intolerance to JNJ-74856665, AZA, or VEN or the excipients of these treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Arms A and D: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 21 Days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Arms B and C: Number of Participants with DLT | Up to 28 Days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Arms A, B, C and D: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | After last dose of study treatment (up to 6 months)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Arms A, B, C and D: Number of Participants with AEs by Severity | After last dose of study treatment (up to 6 months)
  Number of participants with AEs by severity will be reported as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-74856665 | Up to 2 years and 10 months
  Plasma samples will be analyzed to determine concentrations of JNJ-74856665.
Biomarker Levels of Intermediates Including Dihydroorotate (DHO), Orotate, and Uridine of JNJ-74856665 | Up to 2 years and 10 months
  Biomarker levels of intermediates including DHO, orotate, and uridine will be measured by liquid chromatography/mass spectrometry (LC-MS) for JNJ-74856665.
Arm A, Arm B and Arm C: Clinical Response of all Participants with a Primary Disease of Acute Myeloid Leukemia (AML) | Up to 2 years and 10 months
  Clinical response will be assessed per the modified European Leukemia Net (ELN) 2017 recommendations.
Arm A, Arm B and Arm C: Clinical Response of all Participants with a Primary Disease of Myelodysplastic Syndrome (MDS) | Up to 2 years and 10 months
  Clinical response will be assessed per the modified International Working Group 2018 response criteria.
Arm A, Arm B and Arm C: Clinical Response of all Participants with a Primary Disease of chronic myelomonocytic leukemia-2 (CMML-2) | Up to 2 years and 10 months
  Clinical response will be assessed per the modified International Working Group 2018 response criteria.
Arm D: Red Blood Cell-Transfusion Independence (RBC-TI) Rate | Up to 2 years and 10 months
  RBC-TI rate will be reported.
Arm D: Overall Improvement Rate | Up to 2 years and 10 months
  Overall improvement rate is defined as the percentage of participants achieving complete remission, partial remission, or hematologic improvement (HI) according to modified International Working Group (IWG) response criteria.
Arms A, B, C and D: Time to Response (TTR) | Up to 2 years and 10 months
  TTR defined for the responders as the time from the date of first dose of study treatment to the date of initial documentation of a first response as defined in the disease-specific response criteria.
Arms A, B, C and D: Duration of Response (DOR) | Up to 2 years and 10 months
  DOR will be calculated from the date of initial documentation of a response to the date of first documented evidence of relapse, as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first. For participants with disease that has not relapsed and who are alive, data will be censored at the last disease evaluation before the start of any subsequent anticancer therapy.
Arms A, B, C and D: Transfusion Independence (TI) | Up to 2 years and 10 months
  TI is defined as the absence of RBC and platelet transfusions for 8 weeks or longer after starting study treatment for participants with a primary diagnosis of AML or CMML-2, and 16 weeks or longer for participants with a primary diagnosis of MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- France (5):
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire (CHU) de Bordeaux Hopital HautLeveque Centre Francois Magendie, Pessac
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU Tours Hopital Bretonneau, Tours
- South Korea (5):
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (6):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (4):
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - Kings College Hospital, London
  - The Christie Nhs Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency